CLINICAL TRIAL: NCT06605560
Title: Ultrasound-guided Baker Cyst Aspiration Combined With Platelet-rich Plasma Injection in Knee Osteoarthritis: a Randomised Clinical Trial
Brief Title: Baker Cyst Aspiration Combined With Platelet-rich Plasma Injection in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ayhan Aşkın, MD, Professor, MD, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-KAEK-76
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pain; Quality of Life; Baker Cyst; Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Baker Cyst; Platelet Rich Plasma
MeSH Terms: conditions — Pain; Popliteal Cyst; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspiration group (No Intervention): The existing Baker's cyst of patients in this group will be aspirated under ultrasonographic guidance.
- PRP+Aspiration group (Experimental): The existing Baker's cyst of patients in this group will be aspirated under ultrasonography guidance and PRP injection will be administered into the cyst.
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Platelet Rich Plasma — PRP contains a high concentration of platelets obtained by centrifugation of autologous blood. After degranulation of platelets, various growth factors and cytokines are released and accelerate cartilage matrix synthesis, restrain synovial membrane inflammation and promote cartilage healing.
  Arms: PRP+Aspiration group

SUMMARY:
Enlargement of any bursa in or around the popliteal fossa (most commonly the gastrocnemio-semimembranosus (GS) bursa) is called a Baker cyst (BC). Common clinical manifestations of BCs are swelling, mass, pain or stiffness, usually worsening with activity. There may be swelling and tightness or pain behind the knee when walking. However, the majority of these cysts are asymptomatic. They can be detected incidentally in the general population but are more commonly found in patients with osteoarthritis of the knee.

In previous studies, aspiration or corticosteroid treatment was frequently used to treat baker's cysts in patients with osteoarthritis and meniscal or ligamentous injuries. However, there is no previous study in the literature showing the efficacy of PRP injection in baker's cyst. In our study, we aimed to compare the efficacy of cyst aspiration and PRP injection into the cyst on pain, function and cyst size compared to cyst aspiration.

DETAILED DESCRIPTION:
The putative mechanism of BC formation in knee OA is the onset of synovial effusion causing an increase in intra-articular pressure, which in turn causes synovial fluid to be forced through a weakened posteromedial joint capsule towards the GS bursa. Anatomically and clinically it can be classified as a primary or, more often, secondary cyst. If there is a connection between the bursa and the knee joint, the cyst is called secondary. Almost all popliteal cysts in adults are secondary. In 30-50% of cases, there is a connection between the knee joint cavity and the gastrocnemio-semimembranosus bursa. The communication canal is a 15-20 mm transverse slit-like capsular opening adjacent to the proximal postero-lateral margin of the medial femoral condyle. There is a "valve" effect between the bursa and the joint due to the movement of the semitendinosus and gastrocnemius muscles. During flexion, the "valve" opens and synovial fluid under pressure moves towards the bursa; during extension, due to the tension of these muscles, the "valve" closes and fluid is trapped in the bursa. Normally the amount of fluid is small and can be easily reabsorbed, but in OA (mainly active knee osteoarthritis) the amount of fluid increases, leading to fullness and the formation of popliteal cysts. The diagnosis of BC can be supported by a number of imaging modalities, including standard radiographs, arthrography, ultrasonography (US), computed tomography, magnetic resonance and magnetic resonance arthrography. US is an excellent method to evaluate the popliteal fossa, showing high sensitivity and specificity in the diagnosis of BC due to its superficial location and the absence of overlying bony structures.

The treatment approach for Baker's cysts ranges from conservative treatments to interventional procedures and surgery. It should be kept in mind that the majority of cysts are secondary in the treatment approach. For this reason, treatment of the primary pathologies causing Baker's cysts occupies an important place in the treatment approach. Conservative treatment includes lifestyle changes, weight loss, rest, ice compression, bandaging, elevation and ROM exercises. In interventional procedures, the most preferred methods are aspiration of the cyst and corticosteroid injection into the cyst. Surgical interventions can be planned as the last treatment option in recurrent baker's cysts with persistent complaints despite conservative and interventional procedures.

Platelet rich plasma (PRP) injections are one of the most commonly used therapies in the treatment of OA. The mechanism of action of PRP is through growth factors. The main growth factors and growth factor families in PRP used in OA treatment include tissue growth factor-β (TGF-β), insulin growth factor 1 (IGF-1), bone morphogenetic proteins (BMP), platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), fibroblast growth factor (FGF) and hepatocyte growth factor (HGF). TGF-β has been identified as one of the most important factors in cartilage regeneration due to its role in the proliferation and differentiation of chondrocytes. TGF-β induces chondrogenic differentiation of MSCs and also antagonizes the suppressive effects of IL-1, a pro-inflammatory cytokine responsible for stimulating catabolic factors and predisposing intracapsular structures to further degradation. IGF-1 is a key component in cartilage development, promoting chondrocyte mitosis and extracellular matrix synthesis. BMP helps chondrocyte migration and FGF has an important role in cartilage repair. PDGF helps regenerate articular cartilage by increasing chondrocyte proliferation and is involved in all cells of mesenchymal origin. VEGF has been shown to influence vascular structure formation and regeneration and is important in restoring nutrient flow. PRP contains a high concentration of platelets obtained by centrifugation of autologous blood. After degranulation of platelets, various growth factors and cytokines are released and accelerate cartilage matrix synthesis, restrain synovial membrane inflammation and promote cartilage healing. Due to its regenerative effect and anti-inflammatory potential properties, PRP is widely used in musculoskeletal diseases such as rotator cuff tear, lateral epicondylitis, patellar tendinopathy, osteoarthritis. PRP is also preferred in the treatment of androgenic alopecia lichen planoplaris acne scatrices in dermatology, in dentistry, in the treatment of corneal ulcers in ophthalmology and in the clinical applications of various branches and its frequency and range of use is increasing day by day. The effectiveness of PRP in knee osteoarthritis has been demonstrated in various studies. Research on the efficacy of PRP has focused on comparing the effects of intra-articular PRP injections with other injection therapies. In many studies, PRP injections improved functional outcomes compared with HA and placebo controls and appear to be more effective in reducing symptoms and improving quality of life. The effects of PRP are apparently longer lasting and superior compared to intramuscular injection therapies. Comparisons between intra-articular PRP injection versus placebo and HA treatment in mild to moderate knee OA have generally shown higher clinical outcome scores with the use of PRP. In moderate knee OA, functional status and pain improved with at least two injections. In late-stage knee OA, only a single intra-articular PRP injection may be sufficient to provide effective pain relief, thus improving activities of daily living and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade 1-2-3 knee osteoarthritis according to Kellgren Lawrence classification
* Presence of a baker cyst (popliteal cyst) with at least one of the width or length measurements >1 cm (proven by magnetic resonans imaging or muskuloskeletal ultrasound examination)

Exclusion Criteria:

* Patients with grade 4 knee osteoarthritis according to the Kellgren Lawrence classification
* Presence of secondary causes other than gonarthrosis which may lead to the development of a Baker cyst, such as meniscopathy, rheumatic diseases or anterior cruciate ligament damage, etc.
* Long-term use (more than 3 months) of corticosteroid-containing medication
* History of hyaluronic acid injection into the knee within the last 6 months or corticosteroid injection within the last 3 months
* Skin lesions in and around the knee area in the last 7 days
* Current Hb value <12 or platelet value <150,000
* Immunologic or connective tissue disease
* Patients with lateral knee joint space narrowing more than medial
* History of previous knee surgery
* History of pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Change from enrollment in the numeric rating scale for pain | (1) From enrollment to the end of treatment at 6 weeks, (2) From enrollment to the end of treatment at 12 weeks
  The numeric rating scale for pain that is a unidimensional measure of pain intensity in adults, including those with chronic pain.The common format is a horizontal bar or line. Similar to the visual analog scale, the numeric rating scale for pain is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from 0 representing one pain extreme (e.g. "no pain") to 11 representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Change from enrollment in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | (1) From enrollment to the end of treatment at 6 weeks, (2) From enrollment to the end of treatment at 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items); Stiffness (2 items) and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change in cyst dimensions (width x length) | (1) From enrollment to the end of treatment at 6 weeks, (2) From enrollment to the end of treatment at 12 weeks
  The ultrasound (US) probe is held with one hand with the long side perpendicular to the femur. Cyst dimensions in mm are calculated by US with the axis perpendicular to the femur as the width and the axis parallel to the femur as the length. Again, cyst area is measured based on the wall of the cyst with the help of US.

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Aşkın, Professor, Principal Investigator — Izmir Katip Çelebi University
Locations (1):
- Izmir Katip Çelebi University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Raeissadat SA, Rayegani SM, Hassanabadi H, Fathi M, Ghorbani E, Babaee M, Azma K. Knee Osteoarthritis Injection Choices: Platelet- Rich Plasma (PRP) Versus Hyaluronic Acid (A one-year randomized clinical trial). Clin Med Insights Arthritis Musculoskelet Disord. 2015 Jan 7;8:1-8. doi: 10.4137/CMAMD.S17894. eCollection 2015. PMID 25624776
- [Background] Deasy BM, Feduska JM, Payne TR, Li Y, Ambrosio F, Huard J. Effect of VEGF on the regenerative capacity of muscle stem cells in dystrophic skeletal muscle. Mol Ther. 2009 Oct;17(10):1788-98. doi: 10.1038/mt.2009.136. Epub 2009 Jul 14. PMID 19603004
- [Background] Braun HJ, Wasterlain AS, Dragoo JL. The use of PRP in ligament and meniscal healing. Sports Med Arthrosc Rev. 2013 Dec;21(4):206-12. doi: 10.1097/JSA.0000000000000005. PMID 24212368
- [Background] Zhao L, Kaye AD, Abd-Elsayed A. Stem Cells for the Treatment of Knee Osteoarthritis: A Comprehensive Review. Pain Physician. 2018 May;21(3):229-242. PMID 29871367
- [Background] Xie X, Zhang C, Tuan RS. Biology of platelet-rich plasma and its clinical application in cartilage repair. Arthritis Res Ther. 2014 Feb 25;16(1):204. doi: 10.1186/ar4493. PMID 25164150
- [Background] Rauschning W. Popliteal cysts (Baker's cysts) in adults. II. Capsuloplasty with and without a pedicle graft. Acta Orthop Scand. 1980 Jun;51(3):547-55. doi: 10.3109/17453678008990839. PMID 7004054
- [Background] Johnson LL, van Dyk GE, Johnson CA, Bays BM, Gully SM. The popliteal bursa (Baker's cyst): an arthroscopic perspective and the epidemiology. Arthroscopy. 1997 Feb;13(1):66-72. doi: 10.1016/s0749-8063(97)90211-5. PMID 9043606
- [Background] Sansone V, De Ponti A. Arthroscopic treatment of popliteal cyst and associated intra-articular knee disorders in adults. Arthroscopy. 1999 May;15(4):368-72. doi: 10.1016/s0749-8063(99)70053-8. PMID 10355711
- [Background] Handy JR. Popliteal cysts in adults: a review. Semin Arthritis Rheum. 2001 Oct;31(2):108-18. doi: 10.1053/sarh.2001.27659. PMID 11590580